CLINICAL TRIAL: NCT00530699
Title: A Phase I, Open Label, Multi-centre Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD1152 in Japanese Patients With Acute Myeloid Leukaemia.
Brief Title: Safety, Tolerability and PK of AZD1152 in Patients With Relapsed Acute Myeloid Leukaemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, Japan Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1531C00008
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Acute Myeloid Leukaemia
Keywords: Acute Myeloid Leukaemia; Phase 1; AZD1152
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 2-((3-((4-((5-(2-((3-fluorophenyl)amino)-2-oxoethyl)-1H-pyrazol-3-yl)amino)quinazolin-7-yl)oxy)propyl)(ethyl)amino)ethyl dihydrogen phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AZD1152 — intravenous

SUMMARY:
The purpose of this study is to assess safety and tolerability of multiple ascending doses of AZD1152 and to assess effect of AZD1152 on the rate of complete remission in patients with relapsed acute myeloid leukaemia who are not considered to be suitable for standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory AML for which no standard therapies are anticipated to result in durable remission
* Newly diagnosed Acute Myeloid Leukemia who are not considered suitable for other treatments.

Exclusion Criteria:

* Administration of anticancer agents (other than hydroxyurea) within 2 weeks prior to first dose of study drug, and administration of hydroxyurea within 24 hours prior to first dose of study drug
* Participation in any other trial with an investigational product within the previous 30 days.
* Uncontrolled intercurrent illness including, but not limited to, active infection, symptomatic congestive heart failure, cardiac arrhythmia or psychiatric illness/social situations

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of AZD1152 in patients with AML by assessment of AEs, vital signs, ECG parameters, clinical chemistry, haematology (including clotting parameters) and urinalysis | assessed at each visit

SECONDARY OUTCOMES:
To examine the pharmacokinetics of AZD1152 | assessed after dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Paul Stockman, Study Director — AstraZeneca
Locations (7):
- Japan (7):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Yoshida-gun, Fukui
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Maebashi, Gunma
  - Research Site, Isehara, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Chūō, Tokyo